CLINICAL TRIAL: NCT01289158
Title: Combined Malonic and Methylmalonic Aciduria (CMAMMA): Gene Identification and Outcome Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Dr. Nancy Braverman, The Research Institute of the MUHC | McGill University Health Centre
Other Study IDs: 10-131-PED
Record Dates: First submitted 2011-02-02; First posted 2011-02-03 (Estimated); Last update posted 2011-02-08 (Estimated); Status verified 2010-10

CONDITIONS: Malonic Aciduria; Methylmalonic Acidemia
Keywords: malonic and methylmalonic aciduria; malonyl-coenzyme A decarboxylase; MLYCD
MeSH Terms: conditions — Malonic aciduria; Methylmalonic acidemia; Macular dystrophy, corneal type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 1. A 5 cc sample of blood from a vein in EDTA tube for DNA testing
  2. A 5 cc sample of urine sample to measure the levels of MA and MMA
  3. An additional 5 cc (1 tsp) of blood sample will be collected from the parents for DNA testing
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- non-classical CMAMMA, classical CMAMMA

SUMMARY:
The investigators are interested in learning more about the changes found in the condition called "Combined elevation of Malonic and MethylMalonic Acid, or CMAMMA. " Malonic, or MA and MethylMalonic, or MMA, are acids formed from the breakdown of protein under normal conditions. However, in the condition called CMAMMA there is an increase of these acids in the blood and urine, which is not normal.

Some people with high MA and MMA in their blood and urine have a serious disease, starting as a baby or young child that includes heart disease and problems in learning. These people have changes in a special enzyme called Malonyl CoA Decarboxylase (MCD). Other people who have a high level of MA and MMA do not have any obvious illness. The investigators are not sure why they have high levels of MA and MMA and why they are not sick.

The goal of this study is to learn more about why some people have a high level of MA and MMA and to make sure there are no medical problems as a result of these high levels. The investigators also want to find out which gene and enzyme cause the high levels of MA and MMA.

ELIGIBILITY:
Inclusion Criteria:

1. Elevated Malonic and Methylmalonic Acid in blood and urine
2. Any age
3. Any sex
4. Asymptomatic

Exclusion Criteria:

1. Defect in malonyl-coenzyme A decarboxylase (MCD) enzyme
2. History of metabolic acidosis, developmental delay and seizures

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Biochemical Genetics clinics patients with non-classical CMAMMA
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada

REFERENCES:
- See also: The Research Institute of the McGill University Health Centre — http://muhc.ca/research/dashboard